CLINICAL TRIAL: NCT00006165
Title: Cultural-based Diabetes Program for Native Hawaiians
Brief Title: Native Hawaiian Diabetes Intervention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Purpose: Prevention
Other Study IDs: maum (completed); DK 48136
Record Dates: First submitted 2000-08-08; First posted 2000-08-09 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Native Hawaiian; Diabetes Mellitus; Lifestyle Intervention; Family Support; Diabetes Mellitus, at-risk
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

INTERVENTIONS:
Behavioral: 'Ohana (Family) Support Lifestyle Intervention

SUMMARY:
The Native Hawaiian Diabetes Intervention Program is a project focused on determining whether a cultural-based, healthy lifestyles program with family support will have a positive effect on lifestyle behaviors and psychosocial and clinical outcomes. A culturally sensitive, lifestyle intervention program was administered via community peer educators to a population of Native Hawaiians with or at risk for diabetes. The effect of this intervention program on selected outcomes is being compared to a ''standard'' program given to a similar population in a second Native Hawaiian community.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a Native Hawaiian adult 30 years of age or older residing in the research community and have diabetes or at-risk for diabetes.
* Family support member must be 18 years or older and live in the study community and be willing to go through the entire program with the participant as their support person.
* Physician clearance to participate in the program.

Exclusion Criteria:

* Pregnancy

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie K. Mau, M. D., Principal Investigator — University of Hawaii
Locations (1):
- University of Hawaii, John A. Burns School of Medicine, Honolulu, Hawaii, United States

REFERENCES:
- [Background] Gilliland SS, Carter JS, Perez GE, Two Feathers J, Kenui CK, Mau MK. Recommendations for Development and Adaptation of Culturally Competent Community Health Interventions in Minority Populations with Type 2 Diabetes Mellitus. Diabetes Spectrum, 11(3):166-174, 1998.
- [Background] Mau MK, Glanz K Chen R, Crabbe K, Severino R, Grove J, Curb JD, Arakaki RF. Lifestyle Behaviors and Mediating Factors for Behavior Change in Response to a Culturally-Responsive Intervention for Native Hawaiians. Diabetes, 1391A, 1999
- [Background] Mau MK, Grandinetti A, Arakaki RF, Chang HK, Kinney EK, Curb JD. The insulin resistance syndrome in native Hawaiians. Native Hawaiian Health Research (NHHR) Project. Diabetes Care. 1997 Sep;20(9):1376-80. doi: 10.2337/diacare.20.9.1376. PMID 9283783
- [Background] Diabetes mellitus and heart disease risk factors in Hawaiians. The Native Hawaiian Health Research Project, RCMI Program. Hawaii Med J. 1994 Dec;53(12):340-3, 364. No abstract available. PMID 7860292
- [Background] Grandinetti A, Chang HK, Mau MK, Curb JD, Kinney EK, Sagum R, Arakaki RF. Prevalence of glucose intolerance among Native Hawaiians in two rural communities. Native Hawaiian Health Research (NHHR) Project. Diabetes Care. 1998 Apr;21(4):549-54. doi: 10.2337/diacare.21.4.549. PMID 9571341